CLINICAL TRIAL: NCT02027636
Title: UPR-CHA Research Center of Excellence- Supplement
Brief Title: Comparative Effectiveness Research for Eliminating Disparities
Acronym: CERED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Puerto Rico (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-0465/08/10; 3P60MD002261 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2014-01-06 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Depression
Keywords: Depression; Latinos; Mental Health; Disparities
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Engagement and Counseling for Latinos (ECLA-F) (Active Comparator): Patients in this arm (ECLA-F) receive the 6-8 session CBT plus care-management intervention, administered in person.
  Interventions: Behavioral: Engagement and Counseling for Latinos (ECLA-F)
- Engagement and Counseling for Latinos (ECLA-T) (Active Comparator): Patients in this arm received the 6-8 session CBT intervention via telephone.
  Interventions: Behavioral: Engagement and Counseling for Latinos (ECLA-T)
- Usual Care (No Intervention): Patients in this arm receive usual care for depression from their primary care providers, which could include antidepressant prescription or referral to specialty mental health care.

INTERVENTIONS:
Behavioral: Engagement and Counseling for Latinos (ECLA-F) — The Engagement and Counseling for Latinos - Face-to-face (ECLA-F) intervention is a cognitive behavioral therapy (CBT) plus care-management intervention delivered in person. The CBT component consists of 6-8 sessions, delivered by a Master's level clinician, and focusing on self-management techniques, problem-solving, and techniques for managing depression and stress. The care-management component of the intervention consisted of monitoring, assistance in scheduling appointments, and help with transportation. This intervention was identical to the telephone (ECLA-F) intervention, except for the delivery method.
  Arms: Engagement and Counseling for Latinos (ECLA-F)
Behavioral: Engagement and Counseling for Latinos (ECLA-T) — The Engagement and Counseling for Latinos - Telephone (ECLA-T) intervention is a cognitive behavioral therapy (CBT) plus care-management intervention delivered via telephone. The CBT component consists of 6-8 sessions, delivered by a Master's level clinician, and focusing on self-management techniques, problem-solving, and techniques for managing depression and stress. The care-management component of the intervention consisted of monitoring, assistance in scheduling appointments, and technical assistance. This intervention was identical to the face-to-face (ECLA-F) intervention, except for the delivery method.
  Arms: Engagement and Counseling for Latinos (ECLA-T)

SUMMARY:
Our study tested the effectiveness of a combined cognitive behavioral therapy (CBT) and care manager intervention offered either by telephone or face-to-face with depressed Latinos identified in primary care. Eligible patients were randomized after baseline to one of three conditions; 1) ECLA-T (telephone) intervention, 2) ECLA-F (face to face) intervention, and 3) usual care. Usual care was considered care as usual in the participating clinic for a patient screening or depression. The ECLA-T intervention was based on a telephone-plus-care-management intervention that has been shown to be effective in decreasing depressive symptoms and increasing client satisfaction and self-perceived global improvement, as compared to usual care in depressed patients in primary care settings.

DETAILED DESCRIPTION:
Our study tested the effectiveness of a combined cognitive behavioral therapy (CBT) and care manager intervention offered either by telephone or face-to-face with depressed Latinos identified in primary care. The study was conducted at two sites (San Juan, PR and Boston, MA), each of which had multiple clinics. Eligible patients were randomized after baseline to one of three conditions; 1) ECLA-T (telephone) intervention, 2) ECLA-F (face to face) intervention, and 3) usual care. Usual care was considered care as usual in the participating clinic for a patient screening or depression. The ECLA-T intervention was based on a telephone-plus-care-management intervention that has been shown to be effective in decreasing depressive symptoms and increasing client satisfaction and self-perceived global improvement, as compared to usual care in depressed patients in primary care settings.

All participants received a baseline interview assessment prior to randomization. After treatment completion (2 to 3 months from baseline), patients completed an end-of-treatment (EOT) assessment, including repeated assessment of baseline measurements. A 4-month follow-up from baseline was scheduled, which replicated the EOT assessment.

For those patients in the intervention conditions, during each session the clinician used CBT and motivational enhancement strategies to engage the patient in treatment and enhance retention. The CBT intervention was composed of a shortened version of the original CBT intervention, comprised of modules that focus on identifying and correcting negative distortions or cognitions, promote behavioral activation through engaging the patient in pleasant activities, and develop supportive relationships. All sessions were tailored within the structured format considering the patient's needs and always employed a collaborative approach with the patient.

The first four sessions occurred weekly. Every other week the clinician evaluated the patient with the PHQ-9 to determine the level of depressive symptoms. After four sessions, if there was improvement two to four more bi-weekly sessions were scheduled. If there was no or minimal improvement, sessions continued weekly up to a total of 8 sessions for a maximum of 3 months treatment. Cases that showed no improvement or deterioration received more intensive monitoring from the supervising clinicians at both sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they are Latinos, at least 18 years of age, score 10 or more on the PHQ-9 and meet at least one of the essential criteria for Major Depressive Disorder (MDD).

Exclusion Criteria:

* Exclusion criteria include history of psychosis, use of any specialty mental health treatment within the 3 months prior to baseline or an appointment with a mental health provider within the next two months, inability to demonstrate capacity to consent or evidence of suicidal thoughts or ideation as measured by an affirmative response to questions 4 and 5 on the Paykel Suicide Questionnaire).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in Depression Severity at baseline, end of treatment (2-3 months), and 6-month follow-up | Baseline, At each intervention visit (approximately weekly up to end of treatment at 2-3 months), and at 6-month follow-up
  Change in severity of depression symptoms will be assessed using two different measures. The Patient Health Questionnaire-9 (PHQ-9) is a nine item depression screening tool, developed and validated for use in primary care settings. The Hopkins Symptom Checklist-20 (HSCL-20) measures depression symptom severity and distress.

SECONDARY OUTCOMES:
Change in Past 30-day Functioning at baseline, end of treatment (2-3 months), and 6-month follow-up | Baseline, At each intervention visit (approximately weekly up to end of treatment at 2-3 months), and at 6-month follow-up
  Overall functioning over the past 30 days was measured using the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2.0).

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, Ph.D., Principal Investigator — Cambridge Health Alliance; Glorisa Canino, Ph.D., Principal Investigator — University of Puerto Rico
Locations (2):
- Cambridge Health Alliance, Somerville, Massachusetts, United States
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- See also: Project Website — http://www.multiculturalmentalhealth.org/cered.asp